CLINICAL TRIAL: NCT02486263
Title: Pathophysiology of the Aerodigestive Reflex in Infants: GERD Management Trial
Brief Title: Neonatal Gastro-Esophageal Reflux Disease (GERD) Management Trial
Acronym: GMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sudarshan Jadcherla (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Sudarshan Jadcherla, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-00734; R01DK068158 (NIH)
Record Dates: First submitted 2015-06-17; First posted 2015-07-01 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: infant; esophagitis; neonate; GERD
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study (Experimental): Treated with omeprazole. This group of subjects will have prescribed restricted feeding volumes, monitored feeding duration time and positioning restrictions
  Interventions: Other: Study Arm - acid suppression plus feeding bundle
- Conventional (Other): Treated with omeprazole. This group of subjects will receive the current standard treatment for Gastro-esophageal reflux disease (GERD) which includes use of acid suppressive medication with no restrictions of the feeding volume, duration or positioning.
  Interventions: Other: Conventional arm - acid suppression only

INTERVENTIONS:
Other: Study Arm - acid suppression plus feeding bundle — * Omeprazole 0.5-1.5 milligrams/kilogram/dose twice a day (BID)
  * Total fluid volume restriction (120-140 milliliters/kilogram/day)
  * Feeding duration over 30 minutes
  * Infant feeds with right side down
  * Infant is placed on back following feeds
  Arms: Study
Other: Conventional arm - acid suppression only — -Omeprazole 0.5-1.5 milligrams/kilogram/dose twice a day (BID)
  Arms: Conventional

SUMMARY:
The overall purpose of the investigator's study is to evaluate the causes of and treatment for feeding difficulty in infants with Gastro-esophageal Reflux Disease (GERD). New treatments can be possible only if the cause is known. Many infants have GERD and feeding difficulties, such as sucking and swallowing problems, vomiting, or delayed emptying of the stomach. Some of these infants have difficulty in protecting their airway during feeding or during reflux, and as a result can breathe fluid into their lungs or hold their breath. Most GERD treatments are done based on experience, but there is no scientific proof that these methods work for infants. GERD and feeding difficulties can lead to longer hospitalization and more stress for the family.

In this clinical trial, the investigators are developing new methods to help with diagnosis as well as defining better treatment strategies in relieving GERD and GERD complications.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) and its troublesome complications constitute serious diagnostic and management challenges to the development of safe feeding and airway protection strategies among infants convalescing in the neonatal intensive care units; thus contributing to prolonged lengths of stay, recurrent hospitalizations, and death. GERD is frequently diagnosed by inadequate criteria, and the relative risks, benefits and indications of GERD therapies are unclear. Significant gaps in knowledge exist in understanding the complex causal or adaptive aerodigestive protective reflex mechanisms implicated in GERD in infants. The long-term goal is to improve digestive health, nutrition, and infant development through the design of simplified personalized treatment paradigms by better understanding the pathophysiology of aerodigestive reflexes.

The current objective is to conduct a prospective single center randomized blinded controlled trial comparing the short term effects of the investigators innovative feeding strategy bundle (study approach) versus standard feeding approach (conventional approach).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized infants with aerodigestive or GERD symptoms
* Gestational age ≤42 weeks
* Premature infants are eligible at 34 weeks postmenstrual age (PMA)
* Enteral or Oral Fed
* Average daily total feeding volume ≥ 150ml/kg/day
* Room air or supplemental oxygen of ≤1 liter/minute (LPM) and/or ≤ 35% by nasal cannula

Exclusion Criteria:

* Known genetic, metabolic or syndromic disease
* Neurological diseases such as Grade 3 or 4 intraventricular hemorrhage (IVH) or intracranial hemorrhage (ICH) and perinatal asphyxia
* Gastrointestinal malformations and surgical gastrointestinal conditions

Ages: 34 Weeks to 60 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2012-12; Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan R Jadcherla, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital
Locations (1):
- The Research Institute at Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jadcherla SR, Hasenstab KA, Wei L, Osborn EK, Viswanathan S, Gulati IK, Slaughter JL, Di Lorenzo C. Role of feeding strategy bundle with acid-suppressive therapy in infants with esophageal acid reflux exposure: a randomized controlled trial. Pediatr Res. 2021 Feb;89(3):645-652. doi: 10.1038/s41390-020-0932-4. Epub 2020 May 7. PMID 32380509
- [Derived] Sultana Z, Hasenstab KA, Moore RK, Osborn EK, Yildiz VO, Wei L, Slaughter JL, Jadcherla SR. Symptom Scores and pH-Impedance: Secondary Analysis of a Randomized Controlled Trial in Infants Treated for Gastroesophageal Reflux. Gastro Hep Adv. 2022;1(5):869-881. doi: 10.1016/j.gastha.2022.06.004. Epub 2022 Jun 20. PMID 36310566
- [Derived] Jadcherla SR, Hasenstab KA, Gulati IK, Helmick R, Ipek H, Yildiz V, Wei L. Impact of Feeding Strategies With Acid Suppression on Esophageal Reflexes in Human Neonates With Gastroesophageal Reflux Disease: A Single-Blinded Randomized Clinical Trial. Clin Transl Gastroenterol. 2020 Nov;11(11):e00249. doi: 10.14309/ctg.0000000000000249. PMID 33259163

RESULTS

PARTICIPANT FLOW:
Groups:
- Study: Treated with omeprazole. This group of subjects will have prescribed restricted feeding volumes, monitored feeding duration time and positioning restrictions
  Study: -Omeprazole 0.75-1.5 milligrams/kilogram/dose twice a day (BID)
  * Total fluid volume restriction (120-140 milliliters/kilogram/day)
  * Feeding duration over 30 minutes
  * Infant feeds with right side down
  * Infant is placed on back following feeds
Period: Overall Study
Arm/Group | Study | Conventional
Started | 40 | 36
Completed | 37 | 35
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population is the same as the participant assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Study | Conventional | Total
Number analyzed (Participants) | 40 | 36 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 36 | 76
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Chronological age at time of inception
  weeks | 10.7 (4.3) | 11.1 (4.5) | 10.9 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 21 | 18 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 39 | 32 | 71
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 27 | 30 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 40 | 36 | 76

OUTCOME MEASURES:

1. Primary Outcome: CLINICAL OUTCOME OF FEEDING SUCCESS
Description: The primary endpoint is the feeding success defined as achieving full oral feeds (defined as no need for tube feeds to maintain hydration and nutrition) and/or a >/= 6 point decrease from baseline symptom score as described by the Infant-Gastro-Esophageal Reflux Questionnaire-Revised. The minimum score is 0 (no symptoms) and the maximum score is 42 (maximum symptoms). Any total score greater than or equal to 16 is considered abnormal.
Time Frame: Up to 5 weeks after enrollment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study | Conventional
Number analyzed (Participants) | 40 | 36
percentage of participants | 33 [19 to 49] | 44 [28 to 62]
Statistical Analysis 1: Comparison: Study vs Conventional; Test type: Superiority; p = 0.28, Chi-squared — The threshold for statistical significance was <0.05

2. Primary Outcome: MOTILITY OUTCOMES: Presence of Esophageal Peristaltic Reflexes
Description: This is part of Aim 2 of this RCT, which is a mechanistic outcome designed to understand the reasons for the clinical outcome. Presence of peristaltic reflex mechanisms elicited upon esophageal provocation during esophageal manometry were compared within the groups, week-5 vs. week-0. Odds ratios (ORs) with 95% confidence interval (CI) are reported from Generalized Estimation Equation models.
Time Frame: 5 weeks
Population: Participants must have motility evaluations completed at week 0 and week 5 and have PPI washout period prior to week 5 evaluation (49 infants had follow up motility studies at week 5 of whom 40 infants had PPI washout while the other 9 remained on PPI due to parental refusal to stop).
Measure: Number (95% Confidence Interval); unit: odds ratio, week-5 vs. week-0
Groups:
- Study: Treated with omeprazole. This group of subjects will have prescribed restricted feeding volumes, monitored feeding duration time and positioning restrictions
  Study Arm - acid suppression plus feeding bundle: -Omeprazole 0.5-1.5 milligrams/kilogram/dose twice a day (BID)
  * Total fluid volume restriction (120-140 milliliters/kilogram/day)
  * Feeding duration over 30 minutes
  * Infant feeds with right side down
  * Infant is placed on back following feeds
Arm/Group | Study | Conventional
Number analyzed (Participants) | 18 | 22
odds ratio, week-5 vs. week-0 | 0.5 [0.3 to 0.9] | 0.7 [0.4 to 1.0]
Statistical Analysis 1: Comparison: Study vs Conventional; Generalized Estimation Equation (GEE) model was used for the comparison of differences between intervention groups from week 0 to week 5 for peristaltic response frequency; Test type: Superiority; p = 0.99, Generalized Estimation Equation — Used Bonferroni adjustment for multiple comparisons. Threshold for statistical significance was p<0.05; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.6] — Data presented as OR (95% CI) using Generalized Estimation Equation (GEE) model with Conventional as reference

3. Secondary Outcome: CLINICAL OUTCOMES: Growth Outcome Measure
Description: Growth: The investigators will measure and track weight growth velocity during the study period
Time Frame: at 5 weeks
Population: Weight not available for three patients in conventional and one patient in study group at time 2
Measure: Mean (Standard Deviation); unit: grams/day
Arm/Group | Study | Conventional
Number analyzed (Participants) | 37 | 35
grams/day | 27.6 (11.1) | 26.5 (7.2)
Statistical Analysis 1: Comparison: Study vs Conventional; Test type: Superiority — Weight velocity in grams/day; p = 0.64, t-test, 2 sided

4. Secondary Outcome: CLINICAL OUTCOME: Development Outcome Measures
Description: Feeding Milestones: The investigators will track feeding method at 1 year.
Time Frame: Up to 1 year age
Population: Those subjects with follow up data available at 1 year of age
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Conventional
Number analyzed (Participants) | 22 | 22
Participants
  PO | 17 | 20
  Transition (PO + tube) | 4 | 0
  Tube | 1 | 2
Statistical Analysis 1: Comparison: Study vs Conventional; Test type: Superiority; p = 0.11, Chi-squared

5. Secondary Outcome: CLINICAL OUTCOME: Respiratory Outcome Measures
Description: Supplemental oxygen requirement at discharge was recorded for both groups
Time Frame: at discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Conventional
Number analyzed (Participants) | 37 | 35
Participants | 7 | 9
Statistical Analysis 1: Comparison: Study vs Conventional; Test type: Superiority; p = 0.49, Chi-squared — Threshold for statistical significance <0.05

ADVERSE EVENTS:
Time Frame: up to 5 weeks during the study period
Arm/Group | Study | Conventional
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/36
Other Adverse Events (participants affected / at risk) | 0/40 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT02486263/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT02486263/Prot_SAP_001.pdf